CLINICAL TRIAL: NCT03748719
Title: A Single Arm Phase II Trial of Preoperative Stereotactic Body Radiation Therapy (SBRT) for T3a or Gleason Grade Group 4 Prostate Cancer
Brief Title: Single Arm Trial of Preoperative Stereotactic Body Radiation Therapy (SBRT) for T3a or Gleason Grade Group 4 Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual interest
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19670
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
Keywords: High Risk Prostate Cancer; prostate; radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Body Radiation Therapy, followed by Prostatectomy (Experimental): Patients will receive 6 Gy per day of Stereotactic Body Radiation Therapy (SBRT) per day for 5 days, followed by prostatectomy in 3 weeks.
  Interventions: Device: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Device: Stereotactic Body Radiation Therapy (SBRT) — SBRT treatment

SUMMARY:
This study involves Stereotactic Body Radiation Therapy (SBRT) followed by prostatectomy (removal of the prostate). SBRT is a relatively new radiation technique in which a few doses of radiation are delivered to small, well-defined tumors. It has been used effectively in other cancers like lung and liver. The radiation will be given for only 5 days.

The purpose of this study is to compare the effects, good and/or bad, of different doses of SBRT given before prostatectomy.

ELIGIBILITY:
* Histologically proven prostate adenocarcinoma.
* Clinical stage ≤T3a based on digital rectal exam (DRE) and ≤T3a based on MRI (within 3 months); N0-Nx; M0-Mx, or Gleason score 4 + 4. No more than 1 lymph node >1 cm.
* PSA ≤ 50 ng/ml, obtained within 3 months
* Prostate volume: ≤60 cc.
* IPSS score ≤15.
* No previous radiotherapy to the prostate or lower pelvis.
* Lymph node risk of <35% using https://www.mskcc.org/nomograms/prostate/pre_op.
* No prior radical prostatectomy or cryotherapy of the prostate (prior transurethral resection or laser ablation are permitted).
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.
* No history of an invasive malignancy (other than this prostate cancer, or non-metastatic basal or squamous skin cancers) in the last 3 years.
* No androgen deprivation therapy (ADT) can be prescribed prior to or during radiation therapy.
* Participant must be able to have gold fiducial markers placed in the prostate. Note: patients can be enrolled after fiducial markers have been placed, as long as the procedure was done in accordance with the protocol (Section 4.2.2).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Ability to understand and the willingness to sign a written informed consent document.
* Willing to fill out quality of life questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Measure of PSA (Prostate Specific Antigen) | Up to 12 months
  Measure of PSA through treatment. PSA is expected to be undetectable (<0.2 mg/ml) after prostatectomy and radiation therapy.
Number of symptomatic adverse anastomotic events | Up to 12 months
  Number of symptomatic anastomotic events related to pre-operative SBRT.

SECONDARY OUTCOMES:
Mean Catheterization Time | Up to 4 weeks post surgery
  Average time of catheterization following prostatectomy
Mean Hospital Stay | Up to 2 week post surgery
  Average time of hospitalization after prostatectomy
Quality of Life assessment | Baseline, at 2 weeks, 4 weeks, 2 months and every 3 months up to 12 months post surgery
  Quality of Life will be assessed using 2 questionnaires: International Prostate Symptom Score (IPSS) and Sexual Health Inventory for Men (SHIM). The IPSS is an eight question questionnaire of symptoms ranging from 0 "not at all" to 5 "always". The SHIM is a five question questionnaire ranging from 1 "almost never or never" to 5 "almost always or always" to determine erectile dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johnstone, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute